CLINICAL TRIAL: NCT04583150
Title: Evolution of Ovarian Reserve in Severely Obese Women After Bariatric Surgery
Brief Title: Ovarian Reserve and Bariatric Surgery
Acronym: BARIAOVO
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180620
Record Dates: First submitted 2020-02-17; First posted 2020-10-12 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Bariatric Surgery; Obesity; Reproductive Health; Fertility
Keywords: Obesity; Bariatric surgery; Gastric bypass; Sleeve; Fertility; Anti-mullerian hormone; Ovarian reserve
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese women with planned surgery (BS group): Obese women with planned BS procedure in standard care
  Interventions: Procedure: Bariatric surgery
- Obese women with no planned surgery (control group): Obese women matched for age and BMI who did not undergo surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Bariatric surgery : sleeve gastrectomy or Roux-en-Y gastric bypass (RYGB)
  Groups: Obese women with planned surgery (BS group)

SUMMARY:
The expansion of the obesity epidemic is accompanied with an increase in bariatric procedures, in particular in women of reproductive age. Severe obesity has negative effects on fertility and on in vitro fertilization (IVF) outcomes, and the weight loss induced by the bariatric surgery (BS) is believed to reverse the deleterious impact of overweight and obesity on female fertility. However, research is limited to retrospective cohort studies, small case-series and case-control studies. Weight reduction has been shown to improve fecundity and hormonal state of a subgroup of obese patients with polycystic ovary syndrome (PCOS). In this population, recent studies have demonstrated an increase of naturally conceived pregnancies following bariatric surgery. However, these studies have evaluated only short-term evolution of ovarian function and not all studies demonstrated improvements in fertility outcomes after BS. Clearly, more studies are needed regarding the effect of BS on obesity-related infertility, and long-term outcome of ovarian function has to be assessed.

Markers of ovarian reserve, including Follicle Stimulating Hormone (FSH), antral follicle count (AFC), and anti-mullerian hormone (AMH), have been used to counsel patients regarding in their reproductive outcomes. Serum AMH concentrations remain remarkably stable throughout the menstrual cycle, which is a great advantage over other markers of fertility. Various studies have evaluated the association between AMH and body mass index (BMI) but reported contradictory results. Some of them have reported a significant inverse correlation between AMH and BMI, but others found no relationship between AMH and BMI. Scarce and small preliminary studies have been performed to evaluate AMH changes after surgical weight loss and showed a decrease in serum AMH.

DETAILED DESCRIPTION:
Medical files of volunteers obese women consulting an endocrinologist nutritionist or a gynaecologist in each center will be screened and women fitting the inclusion criteria will be proposed to participate in the study. These women will be enrolled and matched with obese women with planned bariatric surgery prospectively. The matching for age (± 1 year) and BMI category (BMI 35-39.9 kg/m², 40-49.9 kg/m² and ≥ 50 kg/m²) of each woman in the surgery group with a control woman will be performed globally, i.e. two matched women could belong to the same center or two different centers.

This is a national prospective multicentre cohort study. Obese women with planned BS, matched for presurgical age and BMI with women with no planned BS.

Subjects with planned bariatric surgery will be recruited in the nutrition departments. All consecutive eligible patients will be considered for inclusion.

Obese women with no planned bariatric surgery will be recruited in the same centers than the corresponding women with planned bariatric surgery, but two matched women can belong to two different centers.

All subjects will be followed 36-42 months according to the delay between inclusion and BS, and AMH levels will be measured at baseline or preoperative time, 12, 24 and 36 months after baseline for controls and after BS for operated women.

ELIGIBILITY:
Inclusion Criteria:

Obese women with planned surgery (BS group)

1. Obese women with an indication of bariatric surgery (BMI ≥ 35 kg/m² with an obesity related comorbidity or BMI ≥ 40 kg/m²)
2. Age 18 to 37 years (inclusion possible until the day before the 37th birthday)
3. No pregnancy project in the next 12 months
4. Signed informed consent
5. Affiliated to The French social security except patient on AME (state medical aid)

Obese women with no planned surgery (control group)

1. Obese women with BMI ≥ 35 kg/m²
2. Age 18 to 37 years (inclusion possible until the day before the 37th birthday)
3. No pregnancy project in the next 12 months
4. Signed informed consent
5. Affiliated to the French social security except patient on AME (state medical aid)
6. Matched for age and BMI category (35-39.9 kg/m², 40-49.9 kg/m² and ≥ 50 kg/m²) with an operated woman
7. No bariatric surgery project in the next 12 months

Exclusion Criteria:

For both groups : Obese women with planned bariatric surgery (BS group) and obese women with no planned surgery (control group):

1. Medical condition known to alter ovarian reserve (previous oophorectomy, ovarian surgery, chemotherapy, pelvis or hypothalamic radiotherapy, known premature ovarian insufficiency …)
2. Contraceptive with antigonadotropic action during the month before inclusion
3. Pregnant or lactating woman
4. HIV infection
5. Previous bariatric surgery
6. Expected follow up less than 3 years
7. Absolute contraindication for bariatric surgery (vital risk, anaesthetic contraindication, non stabilized psychiatric disorder, substance addiction)

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Obese women with planned BS procedure vs. obese women matched for age and BMI without BS procedure.
Sampling Method: Non-Probability Sample
Enrollment: 238 (Estimated)
Dates: Start 2020-12-03 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Compare anti-mullerian hormone (AMH) levels in obese women before bariatric surgery and 12 months after the surgery, and at baseline and 12 months in women who did not undergo surgery | Change from baseline to 12 months after bariatric surgery (bariatric surgery group) or to 12 months after inclusion (control group)
  AMH levels will be measured using the AMH Gen II ELISA (Beckman Coulter, ref A79765) whatever the day of the menstrual cycle

SECONDARY OUTCOMES:
Anti-mullerian hormone (AMH) level evolution | before surgery, 12, 24 and 36 months after BS (bariatric surgery group) and at baseline and 12,24 and 36 months (control group)
  Because AMH level is known to decrease with age and the speed of this evolution is mostly unknown in obese women, the deterioration of ovarian reserve in obese women who undergo surgery will be defined according to the natural evolution of AMH level observed in the control group of obese women without bariatric surgery. In operated women, a deterioration will be defined as a decrease of more than 2 standard deviation of the mean decrease observed in non-operated women.
Body composition | before surgery, 12, 24 and 36 months after BS (bariatric surgery group) and at baseline and 12 months(control group)
  by impedancemetry and/or Dual x-ray absorptiometry (DXA) if possible
Hormonal evaluation of Total testosterone | before surgery, 12, 24 and 36 months after BS (bariatric surgery group) and at baseline and 12, 24 and 36 months (control group)
  Hormonal evaluation is evaluated by measuring Total testosterone (ng/ml) in blood samples
Hormonal evaluation of Sex hormone binding globulin | before surgery, 12, 24 and 36 months after BS (bariatric surgery group) and at baseline and 12, 24 and 36 months (control group)
  Hormonal evaluation is evaluated by measuring Sex hormone binding globulin (SHBG) (mmol/l) in blood samples
Hormonal evaluation of Follicle Stimulating Hormone | before surgery, 12, 24 and 36 months after BS (bariatric surgery group) and at baseline and 12, 24 and 36 months (control group)
  Hormonal evaluation is evaluated by measuring Follicle Stimulating Hormone (FSH) (IU/l) in blood samples
Hormonal evaluation of luteinizing hormone | before surgery, 12, 24 and 36 months after BS (bariatric surgery group) and at baseline and 12, 24 and 36 months (control group)
  Hormonal evaluation is evaluated by measuring , luteinizing hormone (LH) (IU/l) in blood samples
Hormonal evaluation of estradiol | before surgery, 12, 24 and 36 months after BS (bariatric surgery group) and at baseline and 12, 24 and 36 months (control group)
  Hormonal evaluation is evaluated by measuring estradiol (pg/ml) in blood samples
Nutritional status by albumin dosage | before and 12, 24 and 36 months after surgery and at baseline and 12 months in controls
  Nutritional status is evaluated by measuring albumin(g/L) in blood samples
Nutritional status by prealbumin dosage | before and 12, 24 and 36 months after surgery and at baseline and 12 months in controls
  Nutritional status is evaluated by measuring prealbumin(g/L) in blood samples
Nutritional status by heamoglobin dosage | before and 12, 24 and 36 months after surgery and at baseline and 12 months in controls
  Nutritional status is evaluated by measuring hemoglobin(g/L) in blood samples
Nutritional status by vitamin B1 dosage | before and 12, 24 and 36 months after surgery and at baseline and 12 months in controls
  Nutritional status is evaluated by measuring vitamin B1(nmol/L or ng/ml) in blood samples
Nutritional status by vitamin B6 dosage | before and 12, 24 and 36 months after surgery and at baseline and 12 months in controls
  Nutritional status is evaluated by measuring vitamin B6(nmol/L or ng/ml) in blood samples
Nutritional status by vitamin B9 dosage | before and 12, 24 and 36 months after surgery and at baseline and 12 months in controls
  Nutritional status is evaluated by measuring vitamin B9(nmol/l) in blood samples
Nutritional status by vitamin B12 dosage | before and 12, 24 and 36 months after surgery and at baseline and 12 months in controls
  Nutritional status is evaluated by measuring vitamin B12(pg/ml or pmol/L) in blood samples
Nutritional status by vitamin D dosage | before and 12, 24 and 36 months after surgery and at baseline and 12 months in controls
  Nutritional status is evaluated by measuring vitamin D(ng/ml or nmol/L) in blood samples
Nutritional status by vitamin E dosage | before and 12, 24 and 36 months after surgery and at baseline and 12 months in controls
  Nutritional status is evaluated by measuring vitamin E(mg/L or µmol/L) in blood samples
Nutritional status by vitamin A dosage | before and 12, 24 and 36 months after surgery and at baseline and 12 months in controls
  Nutritional status is evaluated by measuring vitamin A(ng/ml or µmol/L) in blood samples
Nutritional status by Parathyroid hormone dosage | before and 12, 24 and 36 months after surgery and at baseline and 12 months in controls
  Nutritional status is evaluated by measuring Parathyroid hormone (PTH) (pmol/L or pg/mL) in blood samples
Nutritional status by calcemia dosage | before and 12, 24 and 36 months after surgery and at baseline and 12 months in controls
  Nutritional status is evaluated by measuring calcemia(mmol/L or mg/L) in blood samples
Nutritional status by ferritin dosage | before and 12, 24 and 36 months after surgery and at baseline and 12 months in controls
  Nutritional status is evaluated by measuring ferritin(µg/L) in blood samples
Nutritional status by transferrin saturation coefficient dosage | before and 12, 24 and 36 months after surgery and at baseline and 12 months in controls
  Nutritional status is evaluated by measuring transferrin saturation coefficient(%) in blood samples
Nutritional status by zinc dosage | before and 12, 24 and 36 months after surgery and at baseline and 12 months in controls
  Nutritional status is evaluated by measuring zinc(mg/L or µmol/L) in blood samples
Nutritional status by selenium dosage | before and 12, 24 and 36 months after surgery and at baseline and 12 months in controls
  Nutritional status is evaluated by measuring selenium(µg/L or µmol/L) in blood samples
Metabolic status by fasting blood glucose dosage | before and 12, 24 and 36 months after surgery and at baseline and 12 months in controls
  Metabolic status is evaluated by measuring fasting blood glucose (mmol/L or g/L ) in blood samples
Metabolic status by insulin dosage | before and 12, 24 and 36 months after surgery and at baseline and 12 months in controls
  Metabolic status is evaluated by measuring insulin(µUI/mL) in blood samples
Metabolic status by HbA1c dosage | before and 12, 24 and 36 months after surgery and at baseline and 12 months in controls
  Metabolic status is evaluated by measuring HbA1c(%) in blood samples
Metabolic status by HDL cholesterol dosage | before and 12, 24 and 36 months after surgery and at baseline and 12 months in controls
  Metabolic status is evaluated by measuring HDL cholesterol(mmol/L or g/L ) in blood samples
Metabolic status by LDL cholesterol dosage | before and 12, 24 and 36 months after surgery and at baseline and 12 months in controls
  Metabolic status is evaluated by measuring LDL cholesterol(mmol/L or g/L ) in blood samples
Metabolic status by Triglycerides dosage | before and 12, 24 and 36 months after surgery and at baseline and 12 months in controls
  Metabolic status is evaluated by measuring Triglycerides(mmol/L or g/L ) in blood samples
Metabolic status by creatinine dosage | before and 12, 24 and 36 months after surgery and at baseline and 12 months in controls
  Metabolic status is evaluated by measuring creatinine(µmol/L or mg/L) in blood samples
Number of pregnancies and time to pregnancy (TTP) | before surgery, 12, 24 and 36 months after BS (bariatric surgery group) and at baseline and 12, 24 and 36 months (control group)
Sexuality score | before surgery, 12, 24 and 36 months after BS (bariatric surgery group) and at baseline and 12,24 and 36 months (control group)
  Female Sexual Function Index scale
Sexuality score | before surgery, 12, 24 and 36 months after BS (bariatric surgery group) and at baseline and 12,24 and 36 months (control group)
  Female Sexual Distress Scale-Revised (sexual quality of life) scale
Ultrasound (US) pelvic sonography with follicular antral count (AFC) | before and at 12, 24 and 36 months after surgery, and at baseline and 12 months in controls

CONTACTS AND LOCATIONS:
Overall Officials: CIANGURA Cécile, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (13):
- France (13):
  - CHU Angers, Angers
  - CHU Clermont Ferrand -Site Gabriel Montpied, Clermont-Ferrand
  - AP-HP - Hôpital Louis Mourier, Colombes
  - CHU Dijon Bourgogne - Hôpital Le Bocage Sud, Dijon
  - CHU Grenoble-CSO Grenoble-Arc Alpin, Grenoble
  - CHRU Lille -Hôpial Claude Huriez, Lille
  - HCL - Hôpital Lyon -Sud, Lyon
  - AP-HM - Hôpital Nord, Marseille
  - CHU Montpellier Hôpital Lapeyronie, Montpellier
  - CHU Nantes - Hôpital Nord Laennec, Nantes
  - AP-HP - Groupe Hospitalier Pitié Salpêtrière, Paris
  - AP-HP - Hôpital Europeen Georges Pompidou, Paris
  - 002 CHU Toulouse -Hôpital Rangueil, Toulouse

IPD SHARING:
Plan to Share IPD: No